CLINICAL TRIAL: NCT06092736
Title: Microvascular Angina Intervention With Compound Danshen Dripping Pill (MAIDS)
Acronym: MAIDS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11671808
Record Dates: First submitted 2023-09-24; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-09

CONDITIONS: Microvascular Angina
Keywords: Coronary Blood Flow Reserve; Microvascular Angina; Compound Danshen Dripping Pill; echocardiography
MeSH Terms: conditions — Microvascular Angina

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compound Danshen Dropping Pills (Experimental): Treatment group: Compound Danshen Dropping Pills (Tianjin Tasly Co., Ltd.), orally after meals, 3 times a day, 20 capsules each time.
  Interventions: Drug: Compound Danshen Dropping Pills
- Placebo (Placebo Comparator): Placebo group: placebo (appearance is the same as Compound Danshen Dropping Pills, main ingredient: starch. Production unit: Tianjin Tasly Co., Ltd.), orally after meals, 3 times a day , 20 capsules each time.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Compound Danshen Dropping Pills — Dosage of Compound Danshen Dropping Pills: 20 capsules each time, 3 times a day, after meals. The follow-up period was 6 months.
  Arms: Compound Danshen Dropping Pills
Drug: Placebo — placebo (appearance is the same as Compound Danshen Dropping Pills, main ingredient: starch. Production unit: Tianjin Tasly Co., Ltd.), orally after meals, 3 times a day , 20 capsules each time.
  Arms: Placebo

SUMMARY:
Coronary microvascular disease (MVD) refers to exertional angina or myocardial ischemia caused by abnormal structure and/or function of precoronary arterioles and arterioles under the action of various pathogenic factors. The symptoms of patients with coronary microvascular disease are mainly exertion-related chest pain episodes.

The basic and clinical researches of the traditional Chinese medicine compound Danshen dropping pills have found that it can improve vascular endothelial function and relieve angina pectoris, and it is widely used in clinical practice.

This is a randomized, double-blind, placebo-controlled, multicenter clinical study of Compound Danshen Dropping Pills and blank control in patients with microvascular angina pectoris.

The experimental drug and control drug of this clinical trial were selected according to the ratio of 1:1 patients were enrolled in the pre-experiment.

After the selected patients signed the informed consent, they were divided into a compound Danshen dripping pill treatment group and a placebo group according to a random, double-blind, placebo-controlled method. Dosage of Compound Danshen Dropping Pills or placebo: 20 capsules each time, 3 times a day, for a total of 6 months. Follow-up was performed every 2 months for a total of 6 months.

Primary study endpoints is the difference of the left anterior descending coronary flow reserve (CFR) measured by ultrasound between the two groups compared with the baseline.

Secondary study endpoint include the Number of angina attacks per week, the time of angina pectoris and the time of ischemic ST segment depression in exercise test.

DETAILED DESCRIPTION:
1. Research Background Coronary microvascular disease (MVD) is a clinical syndrome refers to laboratory evidence of exertional angina or myocardial ischemia caused by structural and/or functional abnormalities of precoronary arterioles and arterioles under the influence of multiple pathogenic factors.. The main symptoms of patients with coronary microvascular disease are exertion-related chest pain attacks. It is difficult to distinguish patients with coronary microvascular disease from patients with severe coronary stenosis based on symptoms alone. However, the following clinical characteristics suggest that patients have coronary microvascular disease. It is more likely. First of all, it is more common in women, accounting for about 56%-79% of patients with coronary microvascular disease. However, most female patients with coronary microvascular disease have their first symptoms after menopause, which is no different from traditional female coronary heart disease patients. Secondly, most of the symptoms are induced by exertion, but it is not uncommon to have patients with silent chest pain. There are fewer patients with coronary microvascular disease who simply present with silent chest pain. Impaired coronary dilatation, increased sympathetic stimulation and sensitivity, and exercise-mediated coronary constriction can lead to the development of coronary microvascular dysfunction and reduced coronary flow reserve. Long-term recurrent angina pectoris attacks affect the patient's quality of life. Patients with significantly reduced coronary blood flow reserve or myocardial perfusion reserve, especially female patients, may have a higher incidence of adverse cardiovascular events.

   Regarding drug treatment, traditional anti-ischemic treatment methods are currently recommended, including β- blockers, calcium ion antagonists and nitrates. If symptoms persist, other drugs include angiotensin-converting enzyme inhibitors, statins, ivabradine , ranolazine , and estrogen drugs. However, there is no specific clinical drug treatment. Basic and clinical studies of the traditional Chinese medicine Compound Danshen Dripping Pill have found that it can improve vascular endothelial function and relieve angina pectoris, and is widely used in clinical practice. However, its effect on coronary reserve function and angina pectoris in coronary microvascular disease needs further clinical research to confirm.
2. Study drug The main drug studied in this study is Compound Danshen Dripping Pill. Compound Danshen Dripping Pills (Compound Danshen Dripping Pills, produced by Tasly Holding Group Co., Ltd.) is a compound traditional Chinese medicine preparation composed of Salvia miltiorrhiza, Panax notoginseng, and Borneol. In 1994, it was approved as a drug for the treatment of coronary heart disease and angina pectoris. It has good clinical efficacy and has It has the characteristics of fast onset, low toxicity, small adverse reactions and high safety.

The active ingredients of compound Danshen dripping pills are water-soluble phenolic acids such as salvia miltiorrhiza and Panax notoginseng saponins. During the preparation process, borneol and auxiliary materials are added, and a highly dispersed solid dispersion is made through a specific process. The active ingredients of the drug have high purity, are evenly dispersed, and can be quickly absorbed through the mucous membrane. The dripping pills have good solid dispersion effect. The principle is to melt the drug ingredients and matrix into a solid solution, and the active ingredients of the drug are in the molecular state or in extremely fine form. The crystalline state is highly uniformly dispersed in the matrix, with fast drug dissolution and higher bioavailability. It can be taken sublingually and can quickly relieve angina pectoris and chest tightness.

Compound Danshen Dripping Pill has achieved a full-process quality control method from medicinal materials, intermediates to preparations (GAP-GEP-GMP) through the multi-factor fingerprint quality control system of compound oral Chinese medicine preparations, further improving the full-process quality control system of Compound Danshen Dripping Pill , after testing and analyzing nearly 200 batches of Compound Salvia Miltiorrhizae Dropping Pills Extract and Compound Salvia Miltiorrhizae Dropping Pills, the similarity is over 90%, and the quality of the products is stable between batches. It has been confirmed through the toxicology study of Compound Danshen Dripping Pill and the clinical use of hundreds of millions of people: it has no toxicity, few adverse reactions, and is safe and reliable for long-term use.

As a Chinese patent medicine for the treatment of stable angina pectoris, Compound Danshen Dripping Pill are included in Category A of the 2018 National Essential Drugs Catalog and the 2019 National Basic Medical Insurance, Work Injury Insurance and Maternity Insurance Drug Catalogue. Under the name of "Compound Danshen Dripping Pill", it has been written into more than 20 national medical guidelines or consensus, 15 of which involve the cardiovascular field, including "Guidelines for Rational Medication in Coronary Heart Disease (2nd Edition)", "Acute Myocardial Medication "Guidelines for the Diagnosis and Treatment of Infarction by Integrated Traditional Chinese and Western Medicine", "Chinese Expert Recommendations on the Clinical Application of Compound Danshen Dripping Pill", "Expert Consensus on the Diagnosis and Treatment of Atherosclerosis by Integrated Traditional Chinese and Western Medicine", etc.

In terms of international evidence-based research, large-sample, randomized, double-blind, placebo-controlled RCT studies were used, and 1,004 patients were included in phase III clinical studies at 127 centers in 9 countries/regions around the world, indicating that the US FDA-Phase III The main clinical efficacy indicators: significantly increase the patient's exercise flat time and improve exercise tolerance. Compared with the increase time of exercise oxygen tolerance of similar drugs, Compound Danshen Dripping Pill has obvious advantages . Secondary efficacy indicators: effectively reduce the number of angina attacks per week and significantly reduce the weekly nitroglycerin dosage.

In terms of domestic evidence-based research: 1011 studies on Compound Danshen Dripping Pill for the treatment of stable angina, 16 Meta-analyses, with a total enrollment of more than 100,000 people; 137 studies on the treatment of peri-PCI/ thrombolysis period , the total number of participants exceeds 10000 ; there are 36 studies on Compound Danshen Dripping Pill improving coronary microcirculation disorders, filling the gap in Western medicine treatment.

Systematic study of Compound Danshen Dripping Pill combined with Western medicine in the treatment of coronary heart disease angina pectoris: 21 articles were included, with a total number of cases of 2229. Compound Danshen Dripping Pill combined with Western medicine can benefit patients with coronary heart disease angina pectoris, especially in improving clinical symptoms and electrocardiogram . It has outstanding effects on ischemic state and regulating cholesterol levels.

A meta-analysis based on PubMed, EMBASE, CNKI, and Wanfang databases studied the efficacy of aspirin combined with Compound Danshen Dripping Pill in the treatment of coronary heart disease. The analysis included 14 randomized controlled trials with a total of 1,367 patients. The results showed that the combination Compared with aspirin alone, the drug can achieve more significant therapeutic effects in relieving angina pectoris symptoms and lowering blood lipids. Lu Yuhong et al. randomly divided 128 patients with coronary heart disease into groups. The control group took oral aspirin on the basis of conventional treatment, and the observation group took Danshen Dropping Pills on the basis of conventional treatment. After 2 months, the total clinical effective rate of the patients in the observation group was significantly higher than Control group. Compared with before treatment, the maximum platelet aggregation rate and thromboxane B2) levels of the two groups of patients were significantly reduced, and the decrease in the observation group was more obvious than that in the control group . The "Guidelines for the Diagnosis and Treatment of Integrated Traditional Chinese and Western Medicine in Acute Myocardial Infarction", led by Academicians Chen Keji, Academician Ge Junbo, and Professor Zhang Minzhou, were formulated in conjunction with experts in the fields of traditional Chinese medicine, Western medicine, integrated traditional Chinese and Western medicine, and methodology across the country. The guideline clearly states that Compound Danshen Dripping Pill are recommended for the treatment of acute myocardial infarction. The recommendation level is the highest in the guideline. Compound Danshen Dripping Pill can relieve chest pain, reduce the patient's risk of cardiac death, and improve the patient's cardiac function. and the role of quality of life.

3. Research purpose A randomized, double-blind, placebo-controlled, multi-center clinical study of Compound Danshen Dripping Pill and blank control was conducted in patients with microvascular angina pectoris .

4. research design 4.1 Study title and registration The Chinese name of this project is: Microvascular Angina Intervention with Compound Danshen Dripping Pill. English name: Microvascular Angina Intervention with Compound Danshen Dripping Pill. Referred to as MAIDS Study.

4.2 Research design : Randomized, double-blind, placebo parallel-controlled, multi-center clinical study.

4. 3 dosing regimens (double-blind single simulation)

1. Placebo group: Placebo (the appearance is the same as Compound Danshen Dripping Pill , main ingredient: starch. Production unit: Tianjin Tasly Co., Ltd.), taken orally after meals, 3 times a day, 20 pills each time .
2. Treatment group: Compound Danshen Dripping Pill (Tianjin Tasly Co., Ltd.), taken orally after meals, 3 times a day, 20 pills each time .

Note: The batch number on the drug packaging is unified as " 161299 ". 5. Research objects 5.1 Source of patients: patients with chest pain who had no obvious coronary artery stenosis on coronary angiography or coronary CT examination were admitted to the hospital outpatient clinics and wards .

5.2Selection criteria _

1. With typical symptoms of exertional angina;
2. Coronary CTA or angiography with normal coronary artery or <50% stenosis, or <50% residual coronary stenosis after revascularization;
3. Ischemic downward shift of the ST segment is found in the electrocardiogram at rest or during exercise stress (horizontal or downsloping downward shift behind the J point >0.1mv, lasting 0.08s );
4. Transthoracic ultrasound before and after intravenous adenosine injection to check the anterior descending coronary artery blood flow reserve test CFR <2.5;
5. The patient agreed to participate in this study. 5.3 Exclusion criteria (1) Aged less than 30 years old or older than 75 years old; (2) Have a history of carotid endarterectomy or stent implantation, and have a history of stroke ; (3) Myocarditis, pericardial disease, valvular disease, and cardiomyopathy; (4) Difficult-to-control diabetes (fasting blood glucose >7.0 mmol/L); ( 5 ) Uncontrollable hypertension (SBP>150 mmHg and/or DBP>90 mmHg); ( 6) Familial hypercholesterolemia; ( 7 ) Takayasu arteritis; ( 8 ) Those who are pregnant or lactating, or those who intend to have a child within one year, or those who have not taken effective contraceptive measures during the childbearing age; ( 9 ) Abnormal liver function (serum GPT level exceeds 3.0 times the upper limit of normal value) or abnormal renal function (serum creatinine level exceeds 2 mg/dl); ( 10 ) Other clinically significant respiratory, digestive, blood, infection, immune, endocrine, neuropsychiatric, tumor diseases, etc., which may cause serious danger to patients; ( 11 ) Take K channel openers and traditional Chinese medicine preparations that activate blood circulation and remove blood stasis to improve microcirculation; (12 ) Those allergic to intra-arterial injection of contrast media, blood, and blood products; (13) Patients who are participating in other clinical studies.

6. Research methods 6.1Sample size The experimental drugs and control drugs in this clinical trial will be selected according to the number of cases in a ratio of 1:1. 100 patients were enrolled in the preliminary experiment .

6.2 Random grouping The randomization method adopts the central randomization method. The central randomization system uses DAS2.1.1 software to generate random numbers (00 1 -100) and drug packaging numbers ( B ZH001-100 ). The random numbers and drug packaging numbers are separated in the system . The researcher passes the Apply to the system to obtain the drug packaging number for the subject. The random number and drug packaging number of the same subject are different, but their corresponding treatment plans are consistent within the system.

6.3 Research process After signing the informed consent form, the selected patients were divided into the Compound Danshen Dripping Pill treatment group and the placebo group according to a random, double-blind, placebo-controlled method. Dosage of Compound Danshen Dripping Pill or placebo: 3 times a day, 20 pills each time, for a total of 6 months . Follow-up visits were conducted every 2 months, and the follow-up period was 6 months in total .

6.4 Screening Phase

1. CTA or CAG examination: Coronary artery CTA or angiography examination shows that the coronary arteries are normal or stenotic <50%, and coronary epicardial vasospasm is excluded;
2. Electrocardiogram: Resting or exercise stress test shows ischemic downward shift of ST segment, horizontal or downward shift behind J point >0.1mv, lasting 0.08s.
3. Laboratory tests: Fasting for more than 6 hours, blood routine, urine routine, fasting blood glucose, alanine aminotransferase, aspartate aminotransferase, troponin, serum creatine phosphokinase, urea nitrogen, creatinine , plasma total cholesterol, triglycerides, hypoglycemia The existing data on density lipoprotein cholesterol, high-density lipoprotein cholesterol, high-sensitivity C-reactive protein, and prothrombin time during the screening phase can no longer be reviewed.
4. Echocardiogram:

After signing the informed consent form, the following inspections will be performed: See Appendix 1 for inspection methods.

1. Routine ultrasound examination: two- dimensional dynamic images of left ventricular parasternal long axis, apical four-chamber, apical two-chamber, apical long axis and left ventricular apex level, papillary muscle level, and mitral valve level short-axis sections. At the same time, pulse wave Doppler was used to obtain the diastolic mitral valve orifice blood flow spectrum, and tissue Doppler was used to obtain the mitral valve annular motion spectrum. See Appendix 1 for details.
2. Acoustic contrast adenosine test: First, observe the distal left anterior descending coronary artery under color Doppler guidance, measure the blood flow velocity with pulsed Doppler ultrasound, and then administer the contrast agent SonoVue (add 8.5ml sterile saline to one bottle ) bolus injection, followed by slowly injecting 5 ml of normal saline over 20 seconds, and measuring the blood flow velocity of the distal left anterior descending coronary artery again . Finally, adenosine 140 µg.kg -1 .min -1 was given for 6 minutes by continuous intravenous micropump injection. During the injection process, the coronary blood flow velocity was monitored. Pulse Doppler ultrasound measured the maximum coronary blood flow velocity in the distal left anterior descending artery. This could be repeated at the same time. Acoustic contrast enhances spectral signals.
3. The adenosine test simultaneously records a 12-lead electrocardiogram.
4. After recording the coronary blood flow in the contrast-enhanced ultrasound examination, the two-dimensional short-axis sections of the left ventricular parasternal long axis, apical four- chamber heart, apical two-chamber heart, apical long axis and left ventricular apex level, papillary muscle level, and mitral valve level were recorded. dynamic images.

6.5 Enrollment and follow-up phase

1. Case grouping 100 patients were selected and randomly divided into Compound Danshen Dripping Pill group and control group, 50 cases each. Compound Danshen Dripping Pill: 20 pills, three times a day; Placebo: 20 pills, three times a day.
2. Follow-up observation Follow-up observations were conducted at 2 months, 4 months, and 6 months after inclusion, including clinical conditions, laboratory examinations, and ultrasound examinations. Safety assessment.

7. Efficacy evaluation 7.1 Main observation indicators Difference in left anterior descending coronary flow reserve (CFR) measured by ultrasound at 6 months compared with baseline.

7.2 Secondary observation indicators

1. Difference in left anterior descending coronary flow reserve (CFR) measured by ultrasound at 2 months and 4 months compared with baseline.
2. Number of angina attacks per week;
3. The time when angina pectoris occurs in exercise test; 4 ) The time when ischemic ST segment depression occurs during exercise testing.

8.Safety assessment Including clinical adverse reactions, laboratory indicators, etc. 9. Adverse event observation and reporting 9.1Definition of Adverse Events Adverse events refer to any adverse medical event that occurs to a patient in this clinical trial from the time the patient signs the informed consent form and is selected to participate in the trial to the last follow-up visit, regardless of whether this event is causally related to the above-mentioned drugs. .

NOTE: An adverse reaction may be any discomfort and unconscious signs (including abnormal laboratory test results), symptoms, or disease (new or worsening) related to the medication.

Events that meet the definition of adverse events include:

* Exacerbation of an existing chronic or intermittent disease, including increased frequency and/or intensity.
* A disease that is newly detected or diagnosed after taking the investigational drug, even though it may have been present before the trial began.
* Signs, symptoms, or clinical sequelae suspected of being caused by an interaction.
* Signs, symptoms or clinical sequelae caused by suspected overdose of the investigational drug or concomitant medication (overdose itself is not an adverse event / serious adverse event).
* " Lack of efficacy " or " failure to achieve the expected pharmacological effect " itself is not reported as an adverse event or serious adverse event. However, signs, symptoms, and/or clinical sequelae due to lack of efficacy will also be reported as adverse events or serious adverse events if they meet the definition of an adverse event or serious adverse event.

Events that do not meet the definition of an adverse event include:

* Medical or surgical procedure (e.g., endoscopy, appendectomy); the event leading up to the procedure is an adverse event.
* Situations in which adverse medical events would not occur (social security and / or admission facilitation).
* There was no worsening of pre-existing diseases or conditions that were present or detected at the start of the trial, only expected day-to-day fluctuations.

  * disease being studied , or the expected progression, signs, or symptoms of the disease being studied. Unless the situation is more serious than expected.

Definition of serious adverse event " serious adverse event " is an adverse event that can occur at any dose and will:

* cause death;
* threatening life; Note: " Life-threatening " means that the subject is in danger of death when the event occurs, not that death could theoretically result if the event were more serious.
* Requires hospitalization or prolonged hospitalization; Note: Typically hospitalization refers to a subject staying in the hospital or emergency room (usually at least overnight) to receive observation and/or treatment that cannot be completed in the doctor's office or outpatient clinic. Complications that occur during hospitalization are considered adverse events. An event is classified as a serious adverse event if the complication prolongs hospitalization or meets the criteria for any other serious adverse event. When it cannot be determined whether " hospitalization " occurred or was necessary, it will be treated as a serious adverse event.

Elective hospitalization that does not worsen a pre-existing condition compared with baseline is not an adverse event.

* Causes disability, or affects the ability to work and live; Note: " Disability " refers to a substantial impairment of an individual's ability to carry out normal life. It does not include discomforts of little clinical significance, such as common headaches, nausea, vomiting, diarrhea, influenza, and accidental trauma (such as sprained ankles), which may affect the quality of daily life but will not constitute a substantial disruption.
* Cause congenital malformations; In other cases, medical or scientific judgment should determine whether adverse event reporting is appropriate. For example, some important medical events may not be immediately life-threatening, leading to death or hospitalization, but may harm subjects or require drug or surgical intervention to avoid the serious adverse events listed above. These events should also be considered serious adverse events, such as invasive or malignant cancer, allergic bronchospasm requiring close monitoring in the emergency room or at home, hematologic cachexia, or convulsions that do not result in hospitalization, drug dependence, or drug abuse.

9.2 Adverse drug reactions Definition: Refers to harmful reactions that occur under normal usage and dosage of qualified drugs and have nothing to do with the purpose of medication.

Causal judgment indicators for adverse reaction judgment:

Item 1 : Is there a reasonable sequence between the time of starting medication and the time when the suspicion appears? Item 2 : Whether the suspected adverse reaction conforms to the known adverse reaction type of the drug; Item 3: Whether the suspected adverse reaction can be explained by the patient's pathological condition, concomitant medications, concomitant therapies, or previous therapies; Item 4 : After stopping the drug or reducing the dose, whether the suspected adverse reactions are reduced or disappeared; Item 5 : Whether the same reaction reappears after using the suspected drug again.

Causality judgment criteria: Judgment based on the order of the above five judgment indicators.

It is up to the investigator to evaluate possible associations between adverse events, trial drugs, and concomitant medications according to the table below.

Adverse reaction cause and effect judgment table

critical result Judgment index Project 1 Project 2 Project 3 Item 4 Item 5 Definitely related + + - + + probably related + + - + ? may be relevant + + ± ± ? suspicious + - ± ± ? Impossibly related + - + - -

Explanation: + Affirmation, - Negation, ± Difficult to affirm or deny,? The situation is unknown.

1.Based on the table above, determine the relationship between the following grade 5 adverse events and the drug.

( 1 ) Definitely related, ( 2 ) Probably related, ( 3 ) Possibly related, ( 4 ) Suspicious, ( 5 ) Impossibly related.

2. The incidence rate of adverse reactions is calculated using the total number of 1 + 2 + 3 + 4 cases as the numerator, and all selected cases that can be evaluated for adverse reactions as the denominator.

9.3Recording of adverse events on the basis of comprehensive consideration of comorbidities and concomitant medications, their relevance to the experiment should be evaluated. The relevance of the drug and documented in detail by the physician.

If an adverse event is discovered, the observing physician can decide whether to terminate the observation based on the condition. Cases of drug discontinuation due to adverse events should be followed up and investigated, and the results should be recorded in detail. If any abnormality in safety test indicators ( blood, urine, stool routine, electrocardiogram, liver function, kidney function ) occurs during or after treatment , the adverse event form should be filled in in a timely manner, reviewed at an appropriate time, and communicated with the subject A comprehensive analysis will be conducted on the onset, treatment, etc. to determine whether it is related to the experimental drug.

9.4 Handling of serious adverse events For any serious adverse events that occur during the trial ( including events requiring hospitalization, prolonged hospitalization, disability, affecting work ability, endangering life or death, causing congenital malformations, etc.) during the clinical trial , the researcher shall immediately respond to the patient's request. In addition to taking emergency measures, the subject must also immediately report to the ethics committee of the National Drug Clinical Trial Institution of Shandong University Qilu Hospital and the main research unit Tianjin Tasly Co., Ltd., the unit responsible for the research. The content of the report of serious adverse events should include: patient's name, random number, length of study participation, start date and stop date of serious adverse events, maximum intensity of serious adverse events, possible relationship between serious adverse events and study drugs, due to serious Whether the adverse event required a change in the study drug, the treatment given to the patient as a result of the serious adverse event, concomitant medications if the serious adverse event occurred, and the outcome of the serious adverse event.

10. Data management and statistical analysis 10.1Data management

1. Establish database: The data administrator establishes an EXCEL database based on the research plan and CRF, and sets up logical verification according to the data verification plan (DVP). Release for use after passing the test.
2. Data entry: Data entry personnel conduct independent double entries and double checks. Inconsistent results will be checked and corrected item by item against the CRF until the results are completely consistent.
3. Data questions and answers: After data entry is completed, the data administrator conducts question screening according to DVP's manual verification plan, opens database access to researchers, and answers questions remotely. The data administrator responds to questions and can issue questions again if necessary until the data is "clean".
4. Database locking: After the main researcher, statistical analysts and data managers jointly sign the "database lock record", the data administrator locks the database.
5. Database submission: The data administrator submits the database to the statistician.

10.2 Statistical analysis data set

1. Full analysis set (FAS): a set of all randomly enrolled cases that used the study drug at least once.
2. Per-protocol set (PPS): It is a data set generated by subjects who are fully compliant with the trial protocol. Compliance includes the treatment received, the availability of primary endpoint measurement, and no major impact on the trial protocol. Violation etc. PPS analysis was used for the primary efficacy outcome measure.
3. Safety Data Set (SS): Actual data that received at least one treatment and had post-treatment safety indicator records. The incidence of adverse reactions was based on the number of SS cases as the denominator.

10.3Statistical methods 9.3.1 Subject distribution analysis

1. List the number of subjects selected and completed the trial, and determine three analysis data sets (FAS, PPS, SS).
2. Conduct a classification analysis on the reasons for not entering PPS and calculate the number of subjects in different categories.
3. Make a detailed list of group classifications, including the reasons for not being included in PPS/FAS/SS.
4. Draw a flow chart of subject distribution. 10.3.2 Demographic data and baseline analysis

Descriptive statistics Demographic information and other baseline characteristic values:

1. Calculate the number of cases, mean, standard deviation, 95%CI, minimum and maximum values for continuous variables.
2. Count and grade data calculation frequency and composition ratio.
3. Inferential statistical results (P values) are listed as descriptive results. 10.3.3 Medication compliance and concomitant medication analysis

<!-- -->

1. Calculate the percentage of subjects with medication compliance in the range of 80%-120%, and use the χ2 test or Fisher's exact probability method to compare differences between groups.
2. Medication exposure, use t test to compare differences between groups.
3. Calculate the percentage of subjects with combined medications, and use the χ2 test or Fisher's exact probability method to compare differences between groups.

10.3.4 Efficacy analysis (1) Analysis of main efficacy indicators FR measured by ultrasound at 6 months and the baseline between the two groups was compared using t test.

(2) Analysis of secondary efficacy indicators FR measured by ultrasound at 2 months and 4 months and the baseline was compared between the two groups using t test;

* For the number of angina attacks per week, t test was used to compare the differences between groups;

  * For the time of occurrence of angina pectoris in exercise test, t test was used to compare the differences between groups;

    * The time when ischemic ST segment downward shift occurs in exercise test, and the t test is used to compare the differences between groups; 10.3.5 Security analysis (1) Calculate the incidence of adverse events/reactions, serious adverse events/reactions, and adverse events/reactions leading to dropout.

      (2) List a detailed list of cases of various adverse events/reactions, serious adverse events/reactions, and adverse events/reactions leading to dropout.

      (3) List the crosstabs of laboratory tests and electrocardiograms before and after medication.

      (4) Descriptive statistics of changes from baseline in laboratory examinations, electrocardiograms, and vital signs, and actual measured values.

      (5) Make a detailed list of abnormal values in laboratory tests, electrocardiograms, and physical examinations.

10.3.6Statistical software

1. Analysis using S PSS software.
2. All statistical tests adopt two-sided tests, and a P value less than or equal to 0.05 will be considered as statistically significant.
3. Detailed statistical methods will be provided in the statistical analysis plan.

ELIGIBILITY:
Inclusion criteria:

1. with typical symptoms of exertional angina;
2. coronary CTA or angiography with normal coronary artery or <50% stenosis, or <50% residual coronary stenosis after revascularization;
3. resting electrocardiogram or During exercise stress, it was found that the ST segment had an ischemic downward shift (the horizontal or downward slope after the J-point shift > 0.1 mv, lasting 0.08 s);
4. Transthoracic ultrasound examination of blood in the anterior descending coronary artery before and after intravenous injection of adenosine Flow reserve check CFR<2.5;
5. The patient himself agrees to participate in this study.

Exclusion criteria

1. Less than 30 years old or more than 75 years old;
2. Have a history of carotid endarterectomy or stent implantation, and have a history of stroke;
3. Myocarditis, pericardial disease, valvular disease, cardiomyopathy;
4. Difficult to control diabetes mellitus (fasting blood glucose>7.0 mmol/L);
5. Uncontrolled hypertension (SBP>150 mmHg and/or DBP>90 mmHg);
6. Familial hypercholesterolemia;
7. Multiple Takayasu arteritis;
8. Those who are pregnant or lactating, or have fertility intention within one year, or have not taken effective contraceptive measures during the childbearing period;
9. Abnormal liver function (the level of serum GPT is 3.0 times higher than the upper limit of normal value) or abnormal renal function (the level of serum creatinine is more than 2 mg/dl);
10. Other respiratory, digestive, blood, infection, immunity, endocrine, neuropsychiatric, tumor diseases with clinical significance that may cause serious danger to patients;
11. Taking traditional Chinese medicine preparations of K channel opener, promoting blood circulation and removing blood stasis to improve microcirculation;
12. Allergies to intra arterial injection of contrast agents, blood and blood products;
13. Patients who are participating in other clinical studies.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-12-18 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
The change of the left anterior descending coronary flow reserve (CFR)measured by echocardiography. | At the end of 6-month follow-up compared to the baseline
  the difference of the left anterior descending coronary flow reserve (CFR) measured by ultrasound between the two groups.

SECONDARY OUTCOMES:
Number of angina attacks per week. | During 6 months of following up.
  The differences in the number of angina attacks between the two groups.
The time of angina pectoris in exercise test. | At the end of 6-month follow-up compared to the baseline.
  The differences in the time of angina pectoris in exercise test between the two groups.
The time of ischemic ST segment depression in exercise test. | At the end of 6-month follow-up compared to the baseline.
  The differences in the time of ischemic ST segment depression in exercise test between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Yun Zhang, PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share the study protocol,statistical Analysis Plan (SAP)and Informed Consent Form (ICF)of this research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The sharing time period is 6 months to 1 year after the data is released.
Access Criteria: Share IPD under the conditions of protecting the privacy of patients and ensuring the safety of all diseases.
  It is necessary to contact the researcher and open the sharing authority after the researcher's consent.

REFERENCES:
- [Background] Mulvagh SL, Rakowski H, Vannan MA, Abdelmoneim SS, Becher H, Bierig SM, Burns PN, Castello R, Coon PD, Hagen ME, Jollis JG, Kimball TR, Kitzman DW, Kronzon I, Labovitz AJ, Lang RM, Mathew J, Moir WS, Nagueh SF, Pearlman AS, Perez JE, Porter TR, Rosenbloom J, Strachan GM, Thanigaraj S, Wei K, Woo A, Yu EH, Zoghbi WA; American Society of Echocardiography. American Society of Echocardiography Consensus Statement on the Clinical Applications of Ultrasonic Contrast Agents in Echocardiography. J Am Soc Echocardiogr. 2008 Nov;21(11):1179-201; quiz 1281. doi: 10.1016/j.echo.2008.09.009. PMID 18992671
- [Background] Porter TR, Abdelmoneim S, Belcik JT, McCulloch ML, Mulvagh SL, Olson JJ, Porcelli C, Tsutsui JM, Wei K. Guidelines for the cardiac sonographer in the performance of contrast echocardiography: a focused update from the American Society of Echocardiography. J Am Soc Echocardiogr. 2014 Aug;27(8):797-810. doi: 10.1016/j.echo.2014.05.011. No abstract available. PMID 25085408
- [Background] Mygind ND, Michelsen MM, Pena A, Frestad D, Dose N, Aziz A, Faber R, Host N, Gustafsson I, Hansen PR, Hansen HS, Bairey Merz CN, Kastrup J, Prescott E. Coronary Microvascular Function and Cardiovascular Risk Factors in Women With Angina Pectoris and No Obstructive Coronary Artery Disease: The iPOWER Study. J Am Heart Assoc. 2016 Mar 15;5(3):e003064. doi: 10.1161/JAHA.115.003064. PMID 27068634
- [Background] Michelsen MM, Pena A, Mygind ND, Frestad D, Gustafsson I, Hansen HS, Kastrup J, Bech J, Host N, Prescott E. Coronary Flow Velocity Reserve Assessed by Transthoracic Doppler: The iPOWER Study: Factors Influencing Feasibility and Quality. J Am Soc Echocardiogr. 2016 Jul;29(7):709-16. doi: 10.1016/j.echo.2016.02.011. Epub 2016 Mar 31. PMID 27038514
- [Background] Prasad M, McBane R, Reriani M, Lerman LO, Lerman A. Coronary endothelial dysfunction is associated with increased risk of venous thromboembolism. Thromb Res. 2016 Mar;139:17-21. doi: 10.1016/j.thromres.2015.12.024. Epub 2015 Dec 29. PMID 26916291
- [Background] Yao GH, Zhang C, Sun FR, Zhang M, Zhao YX, Zhang PF, Zhong L, Ding SF, Chen WQ, Li XN, Zhang Y. Quantification of transmural gradient of blood flow in myocardial ischemia with real-time myocardial contrast echocardiography and dipyridamole stress test. Ultrasound Med Biol. 2008 Jan;34(1):22-30. doi: 10.1016/j.ultrasmedbio.2007.06.019. Epub 2007 Sep 14. PMID 17854984

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/36/NCT06092736/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/36/NCT06092736/ICF_001.pdf